CLINICAL TRIAL: NCT02250755
Title: Comparison of MRI Sequences T1 and T2 * Cerebral Perfusion to Aid in the Diagnosis and Evaluation of Brain Therapeutic Response With Chemotherapy or Targeted Therapy(s) Lesion(s) in Patients Treated and Followed for a Pulmonary Neoplasia
Brief Title: MRI Perfusion on T1 and T2 Brain Lesion(s)
Acronym: METAPERF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012_27; 2012-A01644-39 (Other: ID RCB number, ANSM)
Record Dates: First submitted 2014-06-05; First posted 2014-09-26 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Lung Carcinoma Metastatic to the Brain
Keywords: MRI perfusion; therapeutic response; chemotherapy; brain metastases
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI T1 T2 sequences (Experimental): comparison of perfusion sequences T1 T2 in patients with brain metastase cancer
  Interventions: Other: MRI T1 T2 sequences

INTERVENTIONS:
Other: MRI T1 T2 sequences — MRI

SUMMARY:
This study therefore aims to assess current treatment recommended by scientific societies [ 6-13 ] , brain MRI with injection of contrast for the diagnosis and monitoring of brain metastases . The recommended dose of this examination gadolinium is from 0.1 to 0.3 mmol / kg [ 14 ] . Sequences infusion different from one center to the other made : some use the infusion T1, other infusion T2 * . No recommendation establishes whether it is preferable to use one or the other of these sequences.

No examination is added for the purposes of protocol. Indications for MRI and the number and timing of MRI checks under this protocol are consistent with what is done in practice . The used type of gadolinium and the injected dose will be identical for both sequences infusion . The assessment shall not in any case the contrast but the interpretation of the sequence itself. Special procedures monitoring implemented embodiment correspond to the two sequences instead of infusion (one of T1-weighted and T2 * in the other ) , in the original MRI and MRI of the first control , in order to compare their effectiveness

DETAILED DESCRIPTION:
Eligibility criteria:

* Major Patients
* Addressed MRI for initial assessment of brain metastases
* At a suspicion of one or more brain metastases in the brain scanner routine screening
* Follow for lung cancer histologically documented
* In the Thoracic Oncology Service Professor Lafitte (contact: Dr Cortot)
* To whom treatment with chemotherapy or targeted therapy (including anti-angiogenic) is considered
* Be socially insured

Main Outcomes measures:

Comparing the area under the ROC curve of different parameters evaluated in T1 and T2 * perfusion during the initial assessment for the diagnosis of maximal tumor response evaluated at 1 year

ELIGIBILITY:
Inclusion Criteria:

* Major Patients
* Addressed to MRI for initial assessment of brain metastases
* At a suspicion of one or more brain metastases in the brain scanner routine screening
* Followed for lung cancer histologically documented in the Thoracic Oncology Service of Professor Lafitte (contact: Dr Cortot)
* To whom treatment with chemotherapy or targeted therapy (including anti-angiogenic) is considered
* Be socially insured-

Exclusion Criteria:

* Absolute contraindication to MRI (pacemaker, implantable pacemaker, metallic foreign body intraorbital)
* Patients minors under guardianship / curatorship
* Patients with impaired judgment skills or unable to receive information
* Pregnant Women
* Patients for which lesions are not compatible with lung metastases
* Patients with brain metastases or already known and explored MRI
* Patients for whom treatment by surgical excision of brain metastases is considered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-06; Primary Completion 2015-05 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Comparing different parameters evaluated in T1 and T2 * perfusion | 3 years
  Comparing the area under the ROC curve of different parameters evaluated in T1 and T2 * perfusion during the initial assessment for the diagnosis of maximal tumor

SECONDARY OUTCOMES:
Evaluation tumor response | 1 year
  Comparison of the area under the ROC curve of the change in the first control of the various parameters measured in T1 and T2 * infusion, for the diagnosis of maximum tumor response evaluated at 1 year
Radiological progression-free survival | 1 year
  Comparison of the ability of the two sequences to predict infusion:
Survival without neurological signs | 1 year
  Comparison of the ability of the two sequences to predict infusion:

CONTACTS AND LOCATIONS:
Overall Officials: Xavier LECLERC, Professor, Study Director — CHRU of Lille
Locations (1):
- Hopital Salengro CHRU de Lille, Lille, France